CLINICAL TRIAL: NCT00326235
Title: Effects of Buspirone in Withdrawal From Opiates
Brief Title: Effects of Buspirone in Opiate Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA013264 (NIH)
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-03

CONDITIONS: Heroin Dependence
Keywords: Opioid withdrawal; Buspirone; Methadone taper
MeSH Terms: conditions — Heroin Dependence | interventions — Buspirone

INTERVENTIONS:
Drug: Buspirone

SUMMARY:
Dependence on heroin is a major public health problem because of its association with criminality, law enforcement costs and healthcare costs. Managed withdrawal is a required first step for a long term drug-free treatment of heroin addicts. Methadone and clonidine have been the mainstay of treatment for the relief of heroin withdrawal symptoms but both have limitations. The purpose of this study was to evaluate the efficacy of buspirone in the alleviation of the withdrawal symptoms experienced by heroin addicts when they stop using heroin. Buspirone is a non opiate drug with no abuse potential, no sedating effects and no withdrawal symptoms.

DETAILED DESCRIPTION:
In an attempt to develop a new opiate detoxification approach, the authors assessed the efficacy of buspirone in the treatment of acute heroin withdrawal. Buspirone, a drug interacting with the serotonergic system was selected because there is evidence that a decrease in serotonergic neurotransmission may be involved in opiate withdrawal symptomatology.

Hospitalized heroin addicts were randomized to 4 groups: 1) placebo; 2) methadone; 3) buspirone 30 mg daily; 4) buspirone 45 mg daily. The double-blind trial started in all patients with a 5-day methadone stabilization period ending with a 30 mg dose. This was followed from day 6 through 12 by placebo in group 1 and by a methadone taper in group 2. Because of its delayed action, buspirone was started on day 1 in groups 3 and 4 and was continued, after methadone discontinuation, through day 12. On day 13, drugs and placebo were discontinued and patients observed through day 14. Withdrawal symptoms were assessed with the "Subjective Opiate Withdrawal Scale" (SOWS) and the "Objective Opiate Withdrawal Scale" (OOWS). Participants met with a research assistant daily for 30 minutes while on an inpatient unit. The study did not interfere with the scheduled ward activities. Results so far indicate that the SOWS and OOWS scores were significantly higher in the Placebo group than in the Methadone, Buspirone 30 mg and Buspirone 45 mg groups. There were no significant differences in SOWS or OOWS scores when the Methadone group was compared to each of the two Buspirone groups or when the two Buspirone groups were compared to one another. Thus buspirone, a non opiate drug with no abuse potential, a safe side effect profile and no withdrawal symptoms at doses of 30 and 45 mg, was as effective as a methadone taper in alleviating the withdrawal symptoms of heroin addicts stabilized for 5 days with, and then withdrawn from, methadone. Additional analyses will be performed using data collected in the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled DSM IV diagnostic criteria for opioid dependence
* used heroin daily for at least the prior 6 months with claimed heroin use of at least 2.5g/week
* physical dependence on opiates as determined by history and observation
* admission urine samples demonstrating heroin use
* expressed willingness to participate in a randomized, double-blind, placebo-controlled study for 14 days.

Exclusion Criteria:

* current or past Axis I psychiatric disorder other than opioid dependence
* evidence of significant neurological, gastrointestinal, hepatic, cardiovascular, renal, endocrine or hematologic disease
* seropositive status for the human immunodeficiency virus

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-01; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Laure Buydens-Branchey, M.D., Principal Investigator — VA New York Harbor Healthcare System
Locations (1):
- VA New York Harbor Healthcare System - Brooklyn Campus, Brooklyn, New York, United States

REFERENCES:
- [Result] Buydens-Branchey L, Branchey M, Reel-Brander C. Efficacy of buspirone in the treatment of opioid withdrawal. J Clin Psychopharmacol. 2005 Jun;25(3):230-6. doi: 10.1097/01.jcp.0000162804.38829.97. PMID 15876901